CLINICAL TRIAL: NCT04201171
Title: The Impact of Different CSII and CGM Systems on Metabolic Control and Quality of Life in Children and Adolescents With Type 1 Diabetes. An Observational Study Form the Norwegian Childhood Diabetes Registry (NCDR)
Brief Title: The Impact of Different CSII and CGM Systems on Different Clinical Outcome Variables in Children and Adolescents With Type 1 Diabetes. An Observational Study Form the Norwegian Childhood Diabetes Registry (NCDR)
Status: Completed | Type: Observational
Sponsor: Helse Fonna (Other)
Collaborators: Oslo University Hospital (Other); Helse Vest (Other); University of Bergen (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/1613
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1D; CSII; CGM; diabetic ketoacidosis; hypoglycemia; HRQOL
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Ketoacidosis; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: CSII and CGM — use of CSII as insulin delivery or CGM as glucose monitoring

SUMMARY:
To examine the effect of continuous subcutaneous insulin infusion (CSII) and continuous glucose monitoring (CGM) on metabolic control, in a large population-based nationwide observational study under real life conditions.

All children and adolescents with type 1 diabetes are investigated,using annual data in 2017 from the population-based Norwegian Childhood Diabetes Registry (NCDR). HbA1c, incidence of diabetes ketoacidosis (DKA) and severe hypoglycemia (SH) are evaluated depending on the use of CSII and CGM in a linear mixed-effects and linear regression model adjusted for age, biologic gender and diabetes duration. Health-related quality of Life (HRQOL) is assessed by using the DISABKIDS diabetes specific module (DDM-10), and associations with the use of CSII, CGM, age, gender and diabetes duration are evaluated.

DETAILED DESCRIPTION:
In Norway, all children with diabetes 0-18 years should, due to a recommendation from the national health care authority, receive their diabetes follow-up in a pediatric department. All pediatric departments participate in the NCDR reporting standardized clinical data on their patients to the NCDR, at diabetes onset and annually, until the patients reach 18 years of age. The data completeness of NCDR is high, on individual level 99 % at diabetes onset, and 98 % on the annual examinations in 2016 - 2017.

In addition, HRQOL data were collected in 2017, using the DISABKIDS diabetes specific module (DDM-10). Children 10-17 years with type 1 diabetes were invited to independently fill out the questionnaire regarding their own disease-related quality of life. All parents to children with type 1 diabetes (independent of the child's age) were invited to fill out the same questionnaire, giving a proxy evaluation of their child's quality of life.

ELIGIBILITY:
Inclusion Criteria:

All registered subjects with type 1 diabetes in the 2017 annual cohort of the NCDR

Exclusion Criteria:

None

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Our cohort consists of 2749 patients with type 1 diabetes, 45.5 % females; mean age was 12.9 years (SD 3.9, min 1.7, max 20.2) and mean diabetes duration was 5.3 years (SD 3.7)
Sampling Method: Non-Probability Sample
Enrollment: 2749 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c | measured at annual follow-up in 2017
DKA | registered at annual follow-up in 2017
  diabetic ketoacidosis leading to hospitalization
SH | registered at annual follow-up in 2017
  Severe hypoglycemia
HRQOL | participation connected to annual follow-up in 2017
  health-related quality of life measured with the DISABKIDS diabetes module DDM-10

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Bratke, MD, Principal Investigator — Haugesund Hospital, Fonna Health Trust, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bratke H, Margeirsdottir HD, Assmus J, Njolstad PR, Skrivarhaug T. Does Current Diabetes Technology Improve Metabolic Control? A Cross-Sectional Study on the Use of Insulin Pumps and Continuous Glucose Monitoring Devices in a Nationwide Pediatric Population. Diabetes Ther. 2021 Sep;12(9):2571-2583. doi: 10.1007/s13300-021-01127-6. Epub 2021 Aug 13. PMID 34389930